CLINICAL TRIAL: NCT01336127
Title: Effectiveness of Occupational Therapy in Parkinson's Disease: a Randomized Controlled Trial
Brief Title: Effectiveness Study of Occupational Therapy in Parkinson's Disease
Acronym: OTiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Princess Beatrix Muscle Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W.OR09-29
Record Dates: First submitted 2011-03-17; First posted 2011-04-15 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Parkinson's Disease
Keywords: Occupational Therapy; Parkinson's Disease; Effectiveness; RCT; Activities of daily living; Participation; Caregiver's Burden; Economic evaluation
MeSH Terms: conditions — Parkinson Disease | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- occupational therapy (Experimental): 10 weeks occupational therapy according to a protocol (OTiP protocol) based on the Dutch guidelines of occupational therapy in Parkinson's disease
  Interventions: Behavioral: Occupational Therapy
- No occupational therapy (No Intervention): Patients and their caregivers in the control group will have no occupational therapy intervention until their last measurement has taken place (6 months).

INTERVENTIONS:
Behavioral: Occupational Therapy — Patients in the experimental group will receive 10 weeks (maximum 16 hours) occupational therapy according to a treatment protocol, which is based on the Dutch evidence based guideline for occupational therapy in Parkinson's Disease and refined for this study.
  Arms: occupational therapy

SUMMARY:
The purpose of this study is to determine the effectiveness of occupational therapy in Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a complex disabling condition progressively affecting activities and participation of patients. Occupational Therapy aims to optimise functional performance and engagement in meaningful roles and activities. The lack of scientific evidence for the effectiveness of Occupational Therapy (OT) in Parkinson's Disease (PD) highlights the urgent need for high quality intervention studies. The Dutch clinical practice guideline for OT in PD (2008)offers a good basis for conducting an intervention study. The completed OTiP pilot underscored the feasibility and the need for a large scale trial.

The OTiP study evaluates the effectiveness of OT in improving daily functioning of patients with PD.

ELIGIBILITY:
Inclusion criteria patients:

* Idiopathic Parkinson's Disease
* Indication for referral to occupational therapy
* Home dwelling

Inclusion criteria caregivers

* Available for informal support minimal two times a week to a patient who participates in the study
* Available to take part in the intervention

Exclusion Criteria:

* Not capable of completing the self assessment forms (i.e. due to language problems or severe cognitive problems_MMSE score < 24).
* Co morbidity with symptoms that interfere with actively taking part in the intervention (e.g psychosis, severe heart condition). Or limitations in activities are dominated by the co morbid condition rather than by Parkinson's Disease.
* Current participation in other allied health research (i.e. PARKFIT)
* Having received occupational therapy intervention in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 3 months
  Perceived activity performance. Three months will be the primary analysis. Effects at follow up will be measured at 6 months (see secondary outcome measures)

SECONDARY OUTCOMES:
Perceive Recall Plan Perform Measure (PRPP) | 3 months
  Observational measure. Activity performance patient
Zarit Burden Inventory (ZBI) | 3 months
  Perceived caregiver burden.(caregiver)
Parkinson's Disease Questionnaire 39 (PDQ-39) | 3 months
  Health related Quality of life (Parkinson specific; patient)
Resource utilization questionnaire | 3 months
  For evaluating costs. (patient and caregiver)
Objective Caregiving Burden | 3 months
  Evaluating hours of care (costs). (caregiver)
Activity Card Sort (ACS) | 3 months
  Participation measure:% retained activities.(patient)
The Utrecht Scale for evaluation of Rehabilitation Participation (USER-P)(section III) | 3 months
  Satisfaction with participation (patient)
Becks depression Inventory (BDI) | 3 months
  Mood and Depression. (patient)
Hospital Anxiety and Depression Scale (HADS) | 3 months
  Mood and depression. (caregiver).
The Utrecht Proactive Coping Competence list (UPCC) | 3 months
  Proactive coping skills. (patient and caregiver)
Fatigue Severity Scale (FSS) | 3 months
  Impact of fatigue (patient)
Canadian Occupational Performance Measure (COPM-satisfaction) | 3 months
  Perceived satisfaction with performance. (patient)
Quality of life-overall | 3 months
  One question on rating overall quality of life (VAS scale). (patient and caregiver).
Zarit Burden Inventory (ZBI) | 6 months
  Perceived caregiver burden. (caregiver)
Parkinson's Disease Questionnaire 39 (PDQ-39) | 6 months
  Health related Quality of life (Parkinson specific)
Objective Caregiving Burden | 6 months
  Evaluating hours of care (costs). (caregiver).
Euroqol EQ-5D | 6 months
  Quality of life. Used for patient and caregiver in evaluation of cost effectiveness
Canadian Occupational Performance Measure (COPM) | 6 months
  Perceived performance in activities. Is primary outcome measure at 3 months, but data of 6 months (follow up) wil be used in a secondary analysis and analysis of cost effectiveness.
Canadian Occupational Performance Measure (COPM-satisfaction) | 6 months
  Perceived satisfaction with performance. (patient)
The Utrecht Scale for evaluation of Rehabilitation Participation (USER-P)(section III) | 6 months
  Satisfaction with participation (patient)
Becks depression Inventory (BDI) | 6 months
  Mood and Depression. (patient)
Hospital Anxiety and Depression Scale (HADS) | 6 months
  Mood and depression. (caregiver).
The Utrecht Proactive Coping Competence list (UPCC) | 6 months
  Proactive coping skills. (patient and caregiver)
Fatigue Severity Scale (FSS) | 6 months
  Impact of fatigue (patient)

CONTACTS AND LOCATIONS:
Overall Officials: Marten Munneke, Phd, Principal Investigator — Radboud University Medical Center
Locations (10):
- Netherlands (10):
  - Meander Medisch Centrum, Amersfoort
  - Gelre Ziekenhuizen, Apeldoorn
  - Tergooiziekenhuizen, Blaricum
  - Deventer Ziekenhuis, Deventer
  - St Jansdal, Harderwijk
  - Tergooiziekenhuizen, Hilversum
  - St. Antonius, Utrecht
  - Diakonessenhuis, Zeist
  - Gelre Ziekenhuizen, Zutphen
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Sturkenboom IH, Hendriks JC, Graff MJ, Adang EM, Munneke M, Nijhuis-van der Sanden MW, Bloem BR. Economic evaluation of occupational therapy in Parkinson's disease: A randomized controlled trial. Mov Disord. 2015 Jul;30(8):1059-67. doi: 10.1002/mds.26217. Epub 2015 Apr 8. PMID 25854809
- [Derived] Sturkenboom IH, Graff MJ, Hendriks JC, Veenhuizen Y, Munneke M, Bloem BR, Nijhuis-van der Sanden MW; OTiP study group. Efficacy of occupational therapy for patients with Parkinson's disease: a randomised controlled trial. Lancet Neurol. 2014 Jun;13(6):557-66. doi: 10.1016/S1474-4422(14)70055-9. Epub 2014 Apr 8. PMID 24726066
- [Derived] Sturkenboom IH, Graff MJ, Borm GF, Adang EM, Nijhuis-van der Sanden MW, Bloem BR, Munneke M. Effectiveness of occupational therapy in Parkinson's disease: study protocol for a randomized controlled trial. Trials. 2013 Feb 2;14:34. doi: 10.1186/1745-6215-14-34. PMID 23374761